CLINICAL TRIAL: NCT06431516
Title: Clinical Outcomes of Medical Treatment for Patients With Significant Unprotected Left Main Coronary Artery Disease
Brief Title: LMCA Treatment Outcome
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, GuangMing Tan, Assistant professor, Chinese University of Hong Kong
Other Study IDs: 2023.230
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Left Main Coronary Artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with significant LMCA disease
- normal patient

SUMMARY:
Left main coronary artery (LMCA) is a major branch of coronary artery and supplies a large bulk of myocardium.

Revascularization by either surgical coronary bypass grafting (CABG) or percutaneous coronary intervention (PCI) is recommended for significant unprotected LMCA disease, with CABG being preferred if there is significant involvement in other coronary arteries1,2. CABG has been demonstrated to confer survival benefit over medical therapies patients with LMCA in earlier clinical trials3,4,5. However, these trials were performed before the wide adoption of modern medical therapies such as antiplatelet and statin. Antiplatelet agents, for example, was only used in 32% of all patients in the Coronary Artery Surgery Study3. Modern day medical treatment for stable coronary artery diseases have been shown to be non-inferior to revascularization in both the COURAGE and ISCHEMIA trials6,7. However, patients with LMCA involvement were mostly excluded from both of these studies. In Hong Kong, the average waiting time for an elective CABG for stable patients with LMCA is around 18 months, during which time the patients are treated with modern medical therapies including high-intensity statin and antiplatelet.

DETAILED DESCRIPTION:
Left main coronary artery (LMCA) is a major branch of coronary artery and supplies a large bulk of myocardium.

Revascularization by either surgical coronary bypass grafting (CABG) or percutaneous coronary intervention (PCI) is recommended for significant unprotected LMCA disease, with CABG being preferred if there is significant involvement in other coronary arteries1,2. CABG has been demonstrated to confer survival benefit over medical therapies patients with LMCA in earlier clinical trials3,4,5. However, these trials were performed before the wide adoption of modern medical therapies such as antiplatelet and statin. Antiplatelet agents, for example, was only used in 32% of all patients in the Coronary Artery Surgery Study3. Modern day medical treatment for stable coronary artery diseases have been shown to be non-inferior to revascularization in both the COURAGE and ISCHEMIA trials6,7. However, patients with LMCA involvement were mostly excluded from both of these studies. In Hong Kong, the average waiting time for an elective CABG for stable patients with LMCA is around 18 months, during which time the patients are treated with modern medical therapies including high-intensity statin and antiplatelet.

ELIGIBILITY:
Inclusion Criteria:

* Patients with significant LMCA disease who were on the waitlist for CABG since 1st January 2000 to 31st December 2020.
* The decision for CABG over PCI as a mode of revascularization for the patients on this waitlist were collectively made by the HEART team

Exclusion Criteria:

* patients with co-existing significant valvular heart disease requiring concomitant surgical intervention, and unstable patients in whom urgent surgical intervention was performed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Categorical variables will be presented as numbers and percentages and continuous data as mean and standard deviation. Kaplan-Meier survival curve will be obtained using time to event analysis will be performed for this study, with the time of CABG referral counted as day 0 and the day of CABG counted as the end of follow-up. Multivariate Cox regression analysis will be conducted to delineate the predictors for primary outcomes.
  Potential implications of this study This study will inform us about the mid-term clinical outcomes of modern-day medical therapy in patients with significant LMCA disease. Potential predictors of adverse outcome could be identified through regression analysis. This might help us to identify and expedite CABG arrangement for patients with these risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 4600 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) which is defined as a composite of death of any cause, myocardial infarction (MI), stroke, or urgent revascularization | 1 year
  Major adverse cardiac and cerebrovascular events (MACCE) which is defined as a composite of death of any cause, myocardial infarction (MI), stroke, or urgent revascularization
Death of any cause. | 1 year
  Death of any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided